CLINICAL TRIAL: NCT01127087
Title: A Pilot Study to Evaluate the Safety and Efficacy of Oxazyme (OC4) in Patients With Hyperoxaluria
Brief Title: Oxazyme in Patients With Hyperoxaluria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: OxThera (Industry)
Responsible Party: Principal Investigator, John Lieske, Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-000676
Record Dates: First submitted 2010-05-14; First posted 2010-05-20 (Estimated); Results first posted 2012-12-24 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-11

CONDITIONS: Hyperoxaluria
Keywords: Hyperoxaluria; Oxazyme; oxalate; enteric hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria | interventions — oxalate decarboxylase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RYGB CaOx Stone Formers (Experimental): Subjects with enteric hyperoxaluria after Roux-en-Y Gastric Bypass (RYGB).
  Dosing: 1gm Oxazyme containing approximately 1600 Units OxDC in a sachet administered BID together with lunch and dinner. Subjects were instructed to open the oxazyme sachets and either sprinkle on food or add to a glass of water or fruit juice and consume the contents with a meal twice daily.
  Interventions: Drug: Oxazyme
- Idiopathic Hyperoxaluria CaOx Stone Formers (Experimental): Subjects with idiopathic hyperoxaluria.
  Dosing: 1gm Oxazyme containing approximately 1600 Units OxDC in a sachet administered BID together with lunch and dinner. Subjects were instructed to open the oxazyme sachets and either sprinkle on food or add to a glass of water or fruit juice and consume the contents with a meal twice daily.
  Interventions: Drug: Oxazyme

INTERVENTIONS:
Drug: Oxazyme — Oxazyme (registered trademark) is a non-systemic orally delivered drug composed of recombinant oxalate decarboxylase (OxDC). It is formulated to enzymatically degrade available dietary oxalate prior to its absorption.
  Dosing: 1gm Oxazyme containing approximately 1600 Units OxDC in a sachet administered BID together with lunch and dinner. Subjects were instructed to open the oxazyme sachets and either sprinkle on food or add to a glass of water or fruit juice and consume the contents with a meal twice daily.
  Other Names: oxalate decarboxylase; OC4

SUMMARY:
Hypothesis: Oral administration of the oxalate metabolizing enzyme Oxazyme (OC4) will degrade food-borne oxalate and hence prevent its absorption from the gastrointestinal tract. In addition, by reducing oxalate concentrations in the gastrointestinal fluid, oxalate secretion from blood to the intestinal tract may be increased. Both effects would decrease blood levels of oxalate, and hence oxalate excretion in the urine.

DETAILED DESCRIPTION:
Oxazyme is an oxalate degrading compound that can potentially degrade food-borne oxalate and hence prevent its absorption from the gastrointestinal tract.

We propose a 20-patient open-label trial pilot study of one month of Oxazyme twice daily (1gm Oxazyme sachet dissolved in 150 ml water) among adult subjects with a history of calcium oxalate nephrolithiasis. Patients will be stratified into those with enteric hyperoxaluria after Roux-en-Y Gastric Bypass (RYGB, n=10) and those with idiopathic hyperoxaluria (n=10). The patients will perform two, 24-hour, urine collections immediately before starting Oxazyme and on the last two days of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Roux-en-Y gastric bypass hyperoxaluric Calcium oxalate (CaOx) stone subjects or Idiopathic hyperoxaluric CaOx stone subjects
* Patients must have or had radio-opaque stones present on x-ray, or a history consistent with the passage of a stone or stone surgery or Extracorporeal Shock Wave Lithotripsy (ESWL) in the last 5 years.
* Hyperoxaluria Ox/Cr ratio ≥36 mg/g
* The patient must be able to provide written informed consent
* Patients must be able to urinate reliably into a collection vessel to measure urine volume.
* Patients may be taking drugs for the prevention of stone disease, including pyridoxine, thiazides, citrate supplements and allopurinol, as long as there have been no changes in these medications for at least 3 months

Exclusion Criteria:

* Primary hyperoxaluria patients
* Use of Oxadrop, Oxabsorb, or other therapies affecting oxalate absorption from the gut, other than stable doses of calcium.
* Subjects who are pregnant. Women of childbearing potential must have a negative pregnancy test prior to enrollment and must practice some form of birth control during the trial.
* Patients on an unstable dose of any other drugs for the prevention of stone disease (i.e., pyridoxine, citrate supplements. etc.). Patients should have been on a stable dose for at least 3 months prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lieske, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Mayo Clinic, Rochester, Minnesota.
Pre-assignment Details: 7 subjects were enrolled on the Idiopathic arm; of these 2 did not complete baseline collections, and 3 didn't qualify, so these 5 were excluded. 15 subjects were enrolled on the RYGB arm; of these, 3 never started the study and 2 did not qualify, so these 5 were excluded.
Groups:
- RYGB CaOx Stone Formers: Subjects with enteric hyperoxaluria after Roux-en-Y Gastric Bypass (RYGB).
  Dosing: 1gm Oxazyme containing approximately 1600 Units oxalate decarboxylase (OxDC) in a sachet administered BID together with lunch and dinner. Subjects were instructed to open the oxazyme sachets and either sprinkle on food or add to a glass of water or fruit juice and consume the contents with a meal twice daily.
- Idiopathic Hyperoxaluria CaOx Stone Formers: Subjects with idiopathic hyperoxaluria.
  Dosing: 1gm Oxazyme containing approximately 1600 Units oxalate decarboxylase (OxDC) in a sachet administered BID together with lunch and dinner. Subjects were instructed to open the oxazyme sachets and either sprinkle on food or add to a glass of water or fruit juice and consume the contents with a meal twice daily.
Period: Overall Study
Arm/Group | RYGB CaOx Stone Formers | Idiopathic Hyperoxaluria CaOx Stone Formers
Started | 8 | 2
Completed | 8 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RYGB CaOx Stone Formers | Idiopathic Hyperoxaluria CaOx Stone Formers | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 8
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Urinary Oxalate Creatinine Ratio
Description: The urinary oxalate per creatinine ratio is expressed as mg/g. Paired t-test will be used when comparing reduction of urinary oxalate resulting from treatment (versus baseline) for each subject group.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | RYGB CaOx Stone Formers | Idiopathic Hyperoxaluria CaOx Stone Formers
Number analyzed (Participants) | 8 | 2
mg/g
  Baseline | 68.6 (36.4) | 38.7 (6.9)
  Week 4 | 49.6 (27.9) | 34.7 (6.8)
Statistical Analysis 1: Comparison: RYGB CaOx Stone Formers; Comparison of Urinary oxalate before and at the end of 4 weeks on Oxazyme in the RYGB Calcium oxalate (CaOx) Stone Formers arm; Test type: Superiority or Other; p = 0.027, t-test, 2 sided
Statistical Analysis 2: Comparison: Idiopathic Hyperoxaluria CaOx Stone Formers; Comparison of Urinary oxalate before and at the end of 4 weeks on Oxazyme in the Idiopathic Hyperoxaluria CaOx Stone Formers arm; Test type: Superiority or Other; p = 0.14, t-test, 2 sided

2. Secondary Outcome: Total Urinary Oxalate Excretion
Description: Oxalate is a salt of oxalic acid produced by the body's metabolism and excreted in the urine, measured in this study in two, 24-hour, urine collections.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: mg/24 hrs
Arm/Group | RYGB CaOx Stone Formers | Idiopathic Hyperoxaluria CaOx Stone Formers
Number analyzed (Participants) | 8 | 2
mg/24 hrs
  Baseline | 66.3 (28.0) | 43.2 (5.9)
  4 Weeks | 44.5 (23.7) | 32.3 (3.2)
Statistical Analysis 1: Comparison: RYGB CaOx Stone Formers; Comparison of Oxalate before and at the end of 4 weeks on Oxazyme in the RYGB CaOx Stone Formers arm; Test type: Superiority or Other; p = 0.018, t-test, 2 sided
Statistical Analysis 2: Comparison: Idiopathic Hyperoxaluria CaOx Stone Formers; Comparison of Oxalate before and at the end of 4 weeks on Oxazyme in the Idiopathic Hyperoxaluria CaOx Stone Formers arm; Test type: Superiority or Other; p = 0.06, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The subjects were assessed for adverse events at each site visit and phone follow-up visit.
Arm/Group | RYGB CaOx Stone Formers | Idiopathic Hyperoxaluria CaOx Stone Formers
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 0/8 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No